CLINICAL TRIAL: NCT06037005
Title: The Effect of Cognitive Behavioral Therapy on Post-Traumatic Stress Symptoms in Nursing Students in the COVID 19 Process: Randomized Controlled Trial
Brief Title: The Effect of Cognitive Behavioral Therapy on Post-Traumatic Stress Symptoms in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Fatma Yener Ozcan, Research Assistant, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BDTNurse
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2023-09

CONDITIONS: Trauma and Stressor Related Disorders
Keywords: Nurse; Therapy; Post-Traumatic Stress
MeSH Terms: conditions — Trauma and Stressor Related Disorders

STUDY DESIGN:
Intervention Model Description: Single-blinded study with parallel groups.
Who Masked: Outcomes Assessor
Masking Description: In the study, data collection, statistics and reporting were blinded. The collection of research data and data entry (pre-tests and post-tests and transferring the data to the computer) were carried out by an instructor other than the researcher, who was unaware of the intervention and control groups. Data entries were entered with "A" and "B" codes without specifying the intervention or control group. The analysis of the data and the writing of the research report were coded as "A" and "B" groups. After the statistical analysis was made and the research report was written, the coding for the intervention and control groups was explained to the researcher by the coder.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): Expert support was received from the Cognitive Behavioral Psychotherapy Practitioner and Trainer of the Turkish Psychiatric Association in the creation of the sessions. The researcher applying the therapy has a CBT practitioner certificate. Group intervention program based on cognitive behavioral approach of ten sessions; It was completed in approximately one and a half months (May-June 2022) in the Faculty of Nursing, by dividing the experimental group into two separate groups, two days a week for each group. Each session was held for approximately one hour. The last measurement was made three months after the last therapy session (September 2022).
  Interventions: Other: Cognitive Behavioral Therapy Group
- Control (No Intervention): While group therapy was applied to the experimental group, no intervention was made to the control group.

INTERVENTIONS:
Other: Cognitive Behavioral Therapy Group — Group intervention program based on cognitive behavioral approach of ten sessions; It was completed in approximately one and a half months (May-June 2022) in the Faculty of Nursing, by dividing the experimental group into two separate groups, two days a week for each group. Each session was held for approximately one hour. The last measurement was made three months after the last therapy session (September 2022).
  Arms: Cognitive Behavioral Therapy

SUMMARY:
Objectives: This research was planned to examine the effect of cognitive behavioral therapy on the post-traumatic stress symptoms of nursing students during the COVID-19 pandemic.

Design: Single-blinded study with parallel groups. Setting: Faculty of Nursing. Participants: 60 first-year students studying at the Faculty of Nursing were randomly assigned to the intervention (n=30) and control (n=30) groups.

Method: Data were collected using the Information Form prepared by the researcher and the Post Traumatic Stress Disorder Checklist for DSM-5. The intervention group was collected online three times, before the cognitive behavioral group therapy, at the end of the therapy and three months later. Group intervention program based on cognitive behavioral approach of ten sessions; face-to-face, the intervention group was divided into two separate groups and each group was completed in approximately one and a half months (May-June 2022), two days a week. Follow-up measurement was completed in September 2022. While group therapy was applied to the intervention group, no intervention was made to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being a first year nursing student

Exclusion Criteria:

* Being a foreign student
* Having a psychiatric diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | First assessment will be made at the baseline (pre-intervention)
  Using the Post-Traumatic Stress Disorder Checklist for the DSM-5, symptoms of post-traumatic stress are assessed. Scores ranging from 0 to 80 points are obtained in the scale. In the interpretation of the results of the scale, it gives information about the level of symptoms by calculating the total symptom score together with the sum of the scores of the symptoms in each item, and it is recommended to use 28 as the cut-off point, although it varies according to the purpose of use (Blevins et al., 2015).

SECONDARY OUTCOMES:
Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | The second assessment will take place 5 weeks after the first assessment (after the program is completed).
  Using the Post-Traumatic Stress Disorder Checklist for the DSM-5, symptoms of post-traumatic stress are assessed. Scores ranging from 0 to 80 points are obtained in the scale. In the interpretation of the results of the scale, it gives information about the level of symptoms by calculating the total symptom score together with the sum of the scores of the symptoms in each item, and it is recommended to use 28 as the cut-off point, although it varies according to the purpose of use (Blevins et al., 2015).
Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Third assessment will take place average 12 weeks after the second assessment.
  Using the Post-Traumatic Stress Disorder Checklist for the DSM-5, symptoms of post-traumatic stress are assessed. Scores ranging from 0 to 80 points are obtained in the scale. In the interpretation of the results of the scale, it gives information about the level of symptoms by calculating the total symptom score together with the sum of the scores of the symptoms in each item, and it is recommended to use 28 as the cut-off point, although it varies according to the purpose of use (Blevins et al., 2015).

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Fatma Yener Özcan, Meram, Konya
  - Burcu CEYLAN, Tekirdağ

IPD SHARING:
Plan to Share IPD: No